CLINICAL TRIAL: NCT02090296
Title: Reticulocyte as Risk Marker: Targeted Therapy for Infants With Sickle Cell Anemia
Brief Title: Risk-based Therapy for Sickle Cell Anemia: A Feasibility Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Participant withdrew consent
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Emily Riehm Meier, Attending Physician, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBTSCA
Record Dates: First submitted 2014-02-04; First posted 2014-03-18 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar water (Placebo Comparator): Placebo arm
  Interventions: Other: Placebo
- Hydroxyurea (Active Comparator): Treatment Arm
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea
  Other Names: Hydrea
  Arms: Hydroxyurea
Other: Placebo
  Other Names: Sugar water
  Arms: Sugar water

SUMMARY:
Sickle cell anemia (SCA) patients experience organ damage that begins at an early age and results in significant morbidity and early mortality. Although all SCA patients share the same genetic mutation, the clinical complications are highly variable with some patients experiencing frequent and severe complications, while others have few serious complications. If SCA severity could be predicted early in life, those patients at greatest risk for complications could receive treatment prior to the onset of organ damage. No general SCA severity predictor or one that can be informative early in life exists. The investigators preliminary research has identified the absolute reticulocyte count (ARC) as a potential early predictive risk marker for SCA complications in pediatric patients. A higher ARC between ages 2 and 6 months of age is associated with an increased risk of hospitalization in the first 3 years of life; the mean ARC for the 36 patients who were hospitalized for SCA complications was significantly higher than that of the remaining 23 in those who were not hospitalized. Moreover, total hospitalizations were nearly three times higher by age 2 years in those infants who had an ARC of > 200 than for those infants whose ARC was <200. The proposed study will determine if ARC can be used as a risk-stratifier in asymptomatic infants with SCA and ascertain its value in targeting hydroxyurea therapy to those infants at highest risk of SCA sequelae.

ELIGIBILITY:
Inclusion Criteria:

* ages 6-12 months
* Sickle cell anemia (HbSS)
* steady state absolute reticulocyte count between 2-6 months is available in the medical record

Exclusion Criteria:

* receiving hydroxyurea or chronic monthly blood transfusions
* patient enrolled in preliminary study

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sickle Cell Clinical Change from Baseline to Study Completion ( 18 months) | Every 4 weeks for the 18 months study duration
  Participants will be have a study visit at baseline and then every month for the 18 month duration of the study. Study visits will include a physical exam, laboratory monitoring and interval history to assess the change (if any) every 4 weeks of sickle cell complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States